CLINICAL TRIAL: NCT01911169
Title: Vitamin D Repletion to Improve Endothelial Function in Lupus Patients
Brief Title: Vitamin D to Improve Endothelial Function in SLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jim C. Oates, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00009197
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Atherosclerosis; Systemic Lupus Erythematosus
Keywords: atherosclerosis; systemic lupus erythematosus; flow mediated dilation; interferon gene signature
MeSH Terms: conditions — Atherosclerosis; Lupus Erythematosus, Systemic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D 5000 (Experimental): 5,000 IU vitamin D (cholecalciferol) given orally daily
  Interventions: Drug: Cholecalciferol
- Vitamin D 400 (Active Comparator): cholecalciferol 400 IU daily by mouth
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 5,000 International units versus 400 international units as an active comparator
  Other Names: vitamin D3; Wegman's made by International Vitamin Corporation

SUMMARY:
Determine the effect of vitamin D repletion on flow mediated dilation (FMD, a measure of endothelial function) in vitamin D deficient systemic lupus erythematosus (SLE) patients. The investigators will enroll vitamin D deficient SLE patients and randomize them to receive either 400 IU or 5,000 IU of cholecalciferol (D3) daily and measure change in FMD as a measure of EC function at baseline and after 16 weeks of repletion.

Determine mechanisms by which vitamin D repletion may improve endothelial function in vitamin D deficient SLE patients and in vitro.

Determine effect of oral D3 repletion on the Type I interferon signature in WISH and ECs cultured with pre and post plasma from D3 treated lupus patients.

Determine effect of D3 repletion on the number of circulating apoptotic and non-apoptotic EC and EPC ex vivo.

Determine effect of exogenous 1,25(OH)D on IFN gene signature in WISH and ECs stimulated by pretreatment SLE plasma in vitro.

Determine the effects of exogenous 1,25(OH)D on the phenotype of ECs cultured with pretreatment lupus plasma.

This study is designed to efficiently test our hypothesis and begin to define interferon-dependent pathways through which vitamin D repletion can restore clinical and in vitro endothelial function.

DETAILED DESCRIPTION:
Specific Aim 1. Determine the effect of vitamin D repletion on changes in flow mediated dilation (FMD) in vitamin D deficient SLE patients. The investigators hypothesize that 25(OH)D repletion will improve endothelial function in 25(OH)D deficient lupus patients. For this pilot study, the investigators have opted to use a Randomized Phase II screening design (36). The screening design is meant to provide preliminary comparisons of an experimental treatment to an appropriate control, with the idea that the pilot study would provide valuable information to aid in the design of a definitive Phase III evaluation, should the experimental treatment prove promising in the Phase II trial. The trial is designed to determine the effect of vitamin D repletion with D3 on FMD in vitamin D deficient SLE subjects. Approximately 50 SLE subjects will be screened for total 25(OH) vitamin D (25(OH)D) levels and inclusion/exclusion criteria. However, screening will continue only until 32 participants have been enrolled that have total serum 25(OH)vitamin D levels ≤ 20 ng/ml and meet inclusion/exclusion criteria. A baseline FMD, interferon (IFN) signature assays, and levels of circulating non- and apoptotic endothelial cells (EC) and endothelial progenitor cell (EPC) will be performed at the baseline visit. Participants will be will be randomized into two equal groups of 16 to receive one of two daily oral D3 doses previously used in supplementation trials with no evidence of harm. Group 1 (controls) will receive 400 international units (IU) of D3 daily. Group 2 will receive 5,000 IU daily. Studies of supplementation in subjects deficient in vitamin D demonstrate that supplementation with 1,000, 5,000, and 10,000 IU daily result in increases in 25(OH)D of 4.8, 36.7, and 63.8 ng/mL without evidence of toxicity (37). In this study, steady state levels were achieved at 90 days. As shown in our preliminary studies, 4,000 IU daily is safe and effective at repletion in our lupus clinic population. Some subjects had not achieved steady state at 90 days, so the invesitgators have chosen to dose for 16 weeks. The primary endpoint will be a change in FMD after 16 weeks of vitamin D repletion. The secondary endpoint will be the reduction in IFN signature and level of circulating apoptotic ECs/EPCs in response to vitamin D repletion from baseline to 16 weeks.

Specific Aim 2. Determine mechanisms by which vitamin D repletion may improve endothelial function in vitamin D deficient SLE patients and in vitro.

2.1 Determine effect of oral vitamin D3 repletion on the Type I interferon signature in WISH and ECs cultured with pre and post plasma from D3 treated lupus patients. The investigators hypothesize that the plasma-induced IFN gene signature will reduce with 25(OH)D repletion.

2.2 Determine effect of D3 repletion on the number of circulating apoptotic and non-apoptotic EC and EPC ex vivo. The investigators hypothesize that D3 repletion will reduce the number of apoptotic EC and EPC and increase the number of non-apoptotic EPC in association with improved FMD.

2.3 Determine effect of exogenous 1,25(OH)D on IFN gene signature in WISH and ECs stimulated by pretreatment SLE plasma in vitro. This aim is designed to address the specific question of whether the effect of vitamin D is at least partially due to a direct rather than indirect effect on endothelial response to SLE plasma IFN.

2.4 Determine the effects of exogenous 1,25(OH)D on the phenotype of ECs cultured with pretreatment lupus plasma. This aim was designed to probe the functional significance of vitamin D repletion and reduction of the IFN response on the endothelial phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE per 1997 American College of Rheumatology Criteria(at least 4 criteria present)
* Documented Vitamin D deficiency
* Able to give informed consent

Exclusion Criteria:

* Using tobacco products
* Pregnant/Planning pregnancy
* Known Hypercalcemia (Serum Ca >10.4)
* Known Hypercalcuria (Calcium/Creatinine >0.8)
* Chronic active lupus nephritis or end stage renal disease or kidney stones
* Known Hyperparathyroidism
* Known chronic viral/mycobacterial infections
* Uncontrolled medical disease - Pl judgment
* Current drug or alcohol abuse
* Anticipated poor compliance/known neuropsychiatric disorders
* Hx of cardiovascular events (i.e. Ml, PVD, CVE)
* Subjects taking medications known to affect FMD in lupus subjects such as but not limited to fish oil, statins, will remain on stable doses throughout the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Oates, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Published - 1. Kamen DL, Oates JC.A Pilot Study to Determine if Vitamin D Repletion Improves Endothelial Function in Lupus Patients. Am J Med Sci 2015;350:302-7.
  data available upon request

REFERENCES:
- See also: SCResearch.org is the South Carolina Research Studies Directory designed specifically to help people locate research studies in which to participate. — http://www.scresearch.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initially, subjects will be recruited from the MUSC/UMA clinics. Once interest is confirmed by the subject, study personnel completed a chart review to determine if basic inclusion/exclusion criteria is met. If pre-screen criteria were met, a screening visit was scheduled where the informed consent process will be completed by PI/Sub-I.
Pre-assignment Details: 72 SLE patients were identified with a low 25(OH)D level. Of these, 56 failed further pre-screening based on disease activity, medication use, and known cardiovascular disease. Of the 16 who underwent a screening visit, 7 patients failed to meet criteria for enrollment. Nine patients met inclusion and exclusion criteria and were randomized.
Period: Overall Study
Arm/Group | Vitamin D 5000 | Vitamin D 400
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D 5000 | Vitamin D 400 | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change at Week 16 in % Flow Mediated Dilation in Those Who Did and Did Not Replete Vitamin D
Description: Measures were be performed with a Phillips iU22 Ultrasound system and a L9-3 9 mHz probe in 2D mode by a single operator using EKG gating. Baseline measures of brachial artery diameter will be made after the 10 minutes of rest. The blood pressure cuff, placed on the ipsilateral forearm, was inflated to 50 mmHg above the patient's systolic blood pressure for five minutes and then released. Endothelium-dependent FMD was measured continuously during and for three minutes after cuff release. Subjects rested for 10 minutes. Then, endothelium-independent dilation was measured 3 minutes after administration of 0.4 mg of sublingual nitroglycerine. The outcome (%FMD) was the difference between the average endothelium dependent diameter after cuff deflation and the average baseline diameter. The absolute difference between the % FMD at baseline and 16 week follow up was reported.
Time Frame: from zero to sixteen weeks
Measure: Mean (Standard Deviation); unit: Absolute change in % FMD
Groups:
- Repleted Vitamin D: Participants whose final serum 25(OH) vitamin D was > 32 ng/ml after 16 weeks of oral vitamin D
- Not Repleted Vitamin D: Participants whose vitamin D therapy failed to replete final serum levels to > 32 ng/ml after 16 weeks of treatment
Arm/Group | Repleted Vitamin D | Not Repleted Vitamin D
Number analyzed (Participants) | 6 | 3
Absolute change in % FMD | 1.4 (4.3) | -4.2 (2.7)
Statistical Analysis 1: Comparison: Repleted Vitamin D vs Not Repleted Vitamin D; Effect size of primary outcome was calculated; Test type: Other; Cohen's d = 0.68
Statistical Analysis 2: Comparison: Repleted Vitamin D vs Not Repleted Vitamin D; This study was conducted to determine the effect size for in change in FMD at 16 weeks with 25(OH) therapy. For change in FMD at 16 weeks with 25(OH)D repletion, based on this effect size, to detect significant differences between 2 groups, assuming 1) normally distributed data, 2) the same effect size, 3) alpha= 0.05, and 4) a power of 0.8, 35 patients in each group would be required. Therefore, this was designed as a pilot to determine effect size; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Change in Interferon Signature
Description: This outcome was not measured as planned
Time Frame: from zero to sixteen weeks
Arm/Group | Repleted Vitamin D | Not Repleted Vitamin D
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Vitamin D 5000 | Vitamin D 400
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 1/6 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D 5000 (N=6) | Vitamin D 400 (N=3)
hypotension (Cardiac disorders) | 1 (1) | 0 (0) — one subject who had repletion of vitamin D developed hypotension on her regular anti-hypertensive medication and had to be taken off of anti-hypertensive therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No